CLINICAL TRIAL: NCT04044066
Title: BIomarker-based Prognostic Assessment for Patients With Stable Angina and Acute Coronary Syndromes (BIPass)
Brief Title: Biomarker-based Prognostic Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Peking University Third Hospital (Other); Chinese PLA General Hospital Hospital (Unknown); Peking University First Hospital (Other); Central Hospital of Zibo (Other)
Responsible Party: Sponsor
Other Study IDs: 20172020
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Acute Coronary Syndrome; Stable Angina
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — plasma, whole blood, DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Plasma biomarker — New emerging plasma biomarkers carrying prognositic information

SUMMARY:
Coronary artery disease (including stable angina and acute coronary disease) remains the leading mortality and morbidity worldwide. Improvement in biomarker, imaging research have led to new predictors for the prognosis, which may have great clinical value in the current era of personalized medicine. However, there is no available biomarker-based prediction rule for risk assessment of adverse events in patients with stable angina and acute coronary disease. Therefore, we aim to develop and validate a new biomarker-based risk model to improve the prognostication of adverse events (e.g. ischemic and bleeding events ) in the patient population.

DETAILED DESCRIPTION:
Patients enrolled in Qilu Hospital of Shandong University (Jinan, China), Chinese PLA General Hospital Hospital (Beijing, China) and Peking University First Hospital (Beijing, China) are designed as the development cohort to derive the risk prediction models of ischemic and bleeding events. Patients enrolled in Peking University Third Hospital ( Beijing, China) Zibo Central hospital (Zibo, China) are designed as the independent validation cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients with the diagnosis of any type of coronary artery disease (stable angina, unstable angina, non ST-segment elevation myocardial infarction or ST-segment elevation myocardial infarction)
2. Age ≥18 years of age and <85 years of age
3. Patient or guardian provided informed written consent

Exclusion Criteria:

1. Prior surgery (cardiac or non-cardiac), trauma or clinically evident coagulopathic bleeding (e.g. gastrointestinal, genitourinary, et al)
2. Patient with non-cardiac co-morbidities with life expectancy less than 12 months
3. Patients unwilling or unable to comply with all clinical follow-up schedules at 30 days, 6 months and 12 months after discharge

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this prospective, multicenter registry study, we will consecutively enroll eligible patients according to the pre-specified inclusion and exclusion criteria in 6 tertiary hospitals in China. Patients meeting all eligibility criteria will be tracked and their hospitalization data will be collected including baseline clinical and demographic data, risk factors, blood drawn and storage, lab testing results, angiographic and procedural data (if appropriate), medication and adverse events. Clinical follow-up visits will be sheduled at 30 days, 6 months and 12 months after discharge by telephone contact. Follow-up data will be collected and assessment for death (cardiac, non-cardiac), myocardial infarction, stroke, revascularization or bleeding events will be conducted.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-11-09 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events | 12 months
  a composite of cardiac death, myocardial infarction or stroke
Major bleeding | 12 months
  BARC 3 or more bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang J, Zhang T, Xu F, Gao W, Chen M, Zhu H, Xu J, Yin X, Pang J, Zhang S, Wei M, Chen J, Liu Y, Yu X, Chew DP, Chen Y. GDF-15 at admission predicts cardiovascular death, heart failure, and bleeding outcomes in patients with CAD. ESC Heart Fail. 2023 Oct;10(5):3123-3132. doi: 10.1002/ehf2.14484. Epub 2023 Aug 24. PMID 37620152